CLINICAL TRIAL: NCT02389192
Title: A Phase 1a Open-Label Study to Assess the Safety and Pharmacokinetics of a Single ZMappTM Administration in Healthy Adult Volunteers
Brief Title: Safety and Pharmacokinetics of a Single ZMappTM Administration in Healthy Adult Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 150094; 15-I-0094
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2017-12-27

CONDITIONS: Healthy
Keywords: Ebola; Mono-clonal Antibody
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — ZMapp

ARMS (1):
- OPEN (Experimental): healthy volunteers between the ages of 18-50 to receive a one-time infusion of Zmapp at a dose of 50mg/kg.
  Interventions: Drug: ZMAPP

INTERVENTIONS:
Drug: ZMAPP — ZMappTM, a combination of three mouse/human chimeric monoclonal antibodies (mAbs; c4G6, c2G4, and c13C6-FR1) directed against Ebola virus glycoprotein epitopes

SUMMARY:
Background:

- Ebola is a virus that can spread quickly and causes serious disease. It is currently causing an outbreak in West Africa. There are no approved treatments for Ebola. ZMappTM is a new drug made of natural infection-fighting substances. Researchers want to see if it can treat Ebola.

Objective:

- To assess the safety of ZMappTM and how the body processes it. To measure the immune system response to ZMappTM.

Eligibility:

- Healthy people 18 50 years old.

Design:

* Participants will be screened with a medical history, physical exam, and blood and urine tests. They will have an electrocardiogram (ECG) to measure heart electrical activity. Small pads will be stuck to the arms, legs, and chest.
* Participants will be admitted to the hospital. They will have a physical exam, medication review, and blood samples.
* Two intravenous (IV) lines will be placed into separate arm veins. A needle will be used to guide plastic tubing into the veins. One will be used to take blood samples. The other will be used to give the study drug.
* Participants will be given drugs to help prevent side effects.
* Participants will be given the study drug by IV over 10 12 hours. Participants will be monitored closely and vital signs taken frequently. They may have another ECG.
* Blood samples will be taken before, during, and after the infusion.
* Participants will stay in the hospital 1 or 2 nights after receiving the drug.
* Participants will have several study visits over 90 days after getting the study drug. They will be asked about side effects. They may have a physical exam, and blood may be drawn.

DETAILED DESCRIPTION:
Ebola virus (EBOV) is associated with high morbidity and mortality rates in patients presenting clinical illness. Currently, no agent is approved in the U.S. or elsewhere for the therapeutic treatment of EBOV. The current standard of care for EBOV infection is limited to supportive treatment.

ZMapp TM, a combination of three chimeric human/murine monoclonal antibodies against the EBOV surface glycoprotein found on virions and infected cells, is being developed as a treatment for Ebola virus disease. This is a Phase 1a, open-label study to assess the safety and pharmacokinetics of a single intravenous administration of ZMapp tm in healthy adult volunteers. Three subjects will receive a single intravenous dose of 50mg/kg infusion and be evaluated on study Days 0, 1, 2, 7, 14, 21, 28, 60, and 90. Samples will be collected for pharmacokinetic and immunogenicity assessments at baseline, during, and following infusion. Subjects will be monitored and assessed for safety and the incidence of adverse events over the course of the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adult healthy volunteers 18 to 50 years of age, inclusive.
  2. Able to understand and provide written informed consent.
  3. Body mass index 18 kg/m2 to 29 kg/m2, inclusive, at time of screening.
  4. Female subjects must be of non-childbearing potential (e.g., be confirmed postmenopausal or have undergone surgical sterilization) or must, in conjunction with their sexual partner(s), use a highly effective contraceptive (namely, a long-acting reversible method (IUD, injectable, or implant), or a combination of oral contraception in conjunction with a male condom) during the screening period and for at least 30 days after the infusion of study medication.
  5. Male subjects must either be sterile or agree to use, for the entire duration of the study, a male condom; the female sexual partner must also use a medically acceptable form of birth control (e.g., oral contraceptives), or a highly effective contraceptive (as described in #4 above).
  6. Male subjects must agree to not donate sperm for at least 30 days after the infusion of study medication.

EXCLUSION CRITERIA:

1. Pregnancy or breastfeeding.
2. A positive urine or blood screen for drugs of abuse at time of screening.
3. Prior use of any medical intervention involving antibody products.
4. Active substance abuse or any medical or psychiatric condition that, in the opinion of the principal investigator, could jeopardize the subject's safety or the subject's ability to comply with the protocol requirements.
5. Any chronic medical problem that requires daily medications (except Tylenol, oral contraceptives, vitamins, eye drops, and seasonal allergy medications), or other medical history that in the opinion of the investigator significantly increases the risk associated with a Phase 1 drug.
6. Allergy or intolerance of antihistamines, acetominophen, or catabolic steroids.
7. Active participation in any interventional clinical trial within 6 months prior to the dosing on Day 0 (i.e., received any other investigational drug).
8. Prolonged QTcF interval > 440 ms for males or > 460 ms for females.
9. Other clinically significant ECG abnormality, as determined by the principal investigator.
10. Any clinically significant abnormal hematology, chemistry, coagulation, or urinalysis value, as determined by the principal investigator.
11. Glomerular filtration rate (GFR) of < 80 mL/min, based on the Modification of Diet in Renal Disease equation.
12. Urine-albumin-to-creatinine ratio (UACR) > 30 mg/g.
13. Positive serology for Hepatitis B surface antigen
14. Positive serology for Anti Hepatitis C Antibody
15. Positive ELISA for HIV
16. Known or suspected exposure to Ebola virus.
17. Received investigational vaccine for prevention of EVD.
18. Received investigational treatment for EVD.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03-11; Primary Completion 2017-12-27 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of a single IV infusion of 50 mg/kg of ZMappTM | at 8 time points through 90 days following infusion
To determine serum pharmacokinetics following an intravenous (IV) infusion of 50 mg/kg of ZMappTM | at 8 time points through 90 days following infusion

SECONDARY OUTCOMES:
To assess the development of anti-drug antibodies (ADAs) elicited following a single IV infusion of 50 mg/kg of ZMappTM | at 8 time points through 90 days following infusion

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Davey, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)